CLINICAL TRIAL: NCT01764477
Title: Phase Ib Multicenter, Cohort Dose Escalation Trial to Determine the Safety, Tolerance and Preliminary Antineoplastic Activity of Gemcitabine Administered in Combination With Continuous Intravenous Doses of PRI-724, a CBP/ β- Catenin Inhibitor, to Patients With Advanced or Metastatic Pancreatic Adenocarcinoma Eligible for Second-Line Therapy After Failing First-Line Therapy With FOLFIRINOX (or FOLFOX)
Brief Title: Safety and Efficacy Study of PRI-724 Plus Gemcitabine in Subjects With Advanced or Metastatic Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prism Pharma Co., Ltd. (Industry)
Collaborators: inVentiv Health Clinical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRI-724-102
Record Dates: First submitted 2012-12-12; First posted 2013-01-09 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2015-10

CONDITIONS: Advanced Pancreatic Cancer; Metastatic Pancreatic Cancer; Pancreatic Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — ICG 001

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PRI-724 and Gemcitabine (Experimental): This study will have one arm: all enrolled subjects will be treated with both PRI-724 and Gemcitabine.
  Interventions: Drug: PRI-724

INTERVENTIONS:
Drug: PRI-724 — Gemcitabine: 1000 mg/m2 IV over 30 minutes; once weekly dosing; 3 weeks on with 1 week recovery (4 weeks per cycle)
  PRI-724:
  Cohort 1: 320 mg/m2/day; Cohort 2: 640 mg/m2/day; Cohort 3: 905 mg/m2/day; Continuous IV over 24 hours; daily x 7 days; 1 week on with 1 week recovery × 2 (4 weeks per cycle)

SUMMARY:
Laboratory studies suggest that the study drug may stop cancer cells from growing by affecting an interaction between proteins in the cells referred to as cAMP-response element-binding protein and ß-catenin.

The purpose of this research study is to determine the highest safe dose of study drug that may be used when it is given together with a chemotherapy drug to patients with cancer of the pancreas.

DETAILED DESCRIPTION:
PRI-724 is a small molecule antagonist that binds to the co-activator CBP thereby specifically inhibiting the subset of Wnt/β-catenin-driven genes that are up-regulated in cancer cells. PRI-724 is being developed as a potential antineoplastic agent.

Purpose:

To determine the safety, tolerability, dose-limiting toxicities (DLTs), and maximum tolerated dose (MTD) of sequential escalating doses per cohort of PRI-724 administered in combination with gemcitabine to patients with adenocarcinoma of the pancreas that is locally advanced, metastatic, or otherwise inoperable, who are candidates for second-line therapy after failing first-line therapy with FOLFIRINOX (i.e., folinic acid [leucovorin], fluorouracil, irinotecan, oxaliplatin)

* PRI-724: 320, 640, 905 mg/m2/day, continuous intravenous (CIV) infusion over 24 h, daily × 7 days, 1 week on with 1 week recovery × 2 (4 weeks equals 1 cycle)
* Gemcitabine: 1000 mg/m2 IV over 30 minutes; 3 weeks on with 1 week recovery (4 weeks equals 1 cycle)

Patients with documented, measurable or evaluable adenocarcinoma of the pancreas that is locally advanced, metastatic, or otherwise inoperable, who are candidates for second-line therapy after failing first-line therapy with FOLFIRINOX, will be entered into this phase 1b, multicenter, open-label, non-randomized, dose-escalation per cohort study. The trial is designed to evaluate the safety, tolerability, DLT(s), and MTD of escalating doses of PRI-724, a CBP/ β- catenin inhibitor, when administered in combination with a standard dose of gemcitabine. Correlative studies include characterization of the PK profiles of PRI-724 and gemcitabine, evaluation of the utility of potential PD markers of PRI-724 activity, as well as preliminary assessment of the antineoplastic activity of PRI-724 plus gemcitabine in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, > 18 years of age.
2. Patients with a documented (histologically- or cytologically-proven) epithelial cell/adenocarcinoma of the pancreas that is relapsed, locally advanced, or metastatic.
3. Patients with measurable or evaluable disease according to the response evaluation criteria in solid tumors
4. Patients eligible for second-line therapy after failing first-line therapy with the regimen FOLFIRINOX.
5. Patients with a malignancy that is currently not amenable to surgical intervention, due to either medical contraindications or non-resectability of the tumor.
6. Patients with a Karnofsky Performance Status of 70% to 100% (or equivalent, Eastern Cooperative Oncology Group [ECOG] performance status of 0 or 1); Performance Status Evaluation), and an anticipated life expectancy of ≥ 3 months.
7. Patients, both male and female, who are either not of childbearing potential or who agree to use a medically effective method of contraception during the study and for 3 months after the last dose of study drug.
8. Patients with the ability to understand and give written informed consent for participation in this trial, including all evaluations and procedures as specified by this protocol.

Exclusion Criteria:

1. Women who are pregnant or lactating. Women of child-bearing potential (WOCBP) and fertile men with a WOCBP partner, not using adequate birth control.
2. Patients with islet cell tumors or other non-epithelial cell malignancies of the pancreas.
3. Patients with known CNS (or leptomeningeal) metastases not controlled by prior surgery or radiotherapy, or patients with symptoms suggesting CNS involvement for which treatment is required.
4. Patients with an active second malignancy within the last 2 years with the exception of:

   * Treated, non-melanoma skin cancers
   * Treated CIS of the breast or cervix
   * Controlled, superficial bladder carcinoma
   * T1a or b prostate carcinoma involving < 5% of resected tissue and PSA within normal limits (WNL) since resection
5. Patients with any of the following hematologic abnormalities at baseline:

   * Hemoglobin < 9.0 g/dL
   * Absolute neutrophil count (ANC) < 1,500 per mm3
   * Platelet count < 100,000 per mm3
6. Patients with any of the following serum chemistry abnormalities at baseline:

   * Total bilirubin > 1.5× the ULN for the institution, unless considered due to Gilbert's Syndrome
   * AST or ALT > 3× the ULN for the institution (> 5× ULN if due to hepatic involvement by tumor)
   * Serum albumin < 2.5 g/dL
   * Serum creatinine > 1.5× ULN (or a calculated creatinine clearance < 60 mL/min/1.73 m2)
7. Patients with a significant cardiovascular disease or condition, including:

   * Congestive heart failure (CHF) currently requiring therapy
   * Need for anti-arrhythmic therapy for a ventricular arrhythmias
   * Severe conduction disturbances
   * Angina pectoris requiring therapy
   * Left ventricular ejection fraction (LVEF) < 50% by MUGA or echocardiogram
   * QTcF interval > 450 msec (males) or > 470 msec (females)
   * Uncontrolled hypertension (per Investigator's discretion)
   * Class III or IV cardiovascular disease according to the New York Heart Association's (NYHA) Functional Criteria.
   * Myocardial infarction (MI) within 6 months prior to first study drug administration
8. Patients with known osteopenia or osteoporosis.
9. Patients with a known or suspected hypersensitivity to either gemcitabine or any of the components of PRI-724.
10. Patients with a history of human immunodeficiency virus (HIV) or active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV).
11. Patients with any other serious/active/uncontrolled infection, any infection requiring parenteral antibiotics, or unexplained fever > 38ºC within 2 weeks prior to first study drug administration.
12. Patients with inadequate recovery from acute toxicity associated with any prior antineoplastic therapy
13. Patients with inadequate recovery from any prior surgical procedure, or patients having undergone any major surgical procedure within 1 month prior to first study drug administration.
14. Patients with any other life-threatening illness, significant organ system dysfunction, or clinically significant laboratory abnormality, which, in the opinion of the Investigator, would either compromise the patient's safety or interfere with evaluation of the safety of the study drug
15. Patients with a psychiatric disorder or altered mental status that would preclude understanding of the informed consent process and/or completion of the necessary studies
16. Patients with the inability, in the opinion of the Investigator, to comply with the protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The Maximum Tolerated Dose (MTD) of PRI-724 + Gemcitabine measured by the number of dose limiting toxicities (DLTs) that occur. | 18 months. DLTs will be measured as they occur throughout the patients' time on study.
  If no DLT occurs in the first 3 patients of a cohort, the dose will be escalated to the next dose cohort. If 1 DLT occurs in the first 3 patients of a cohort, that cohort is expanded to 6 patients. If more than 1 DLT occurs in a 6 patient cohort, escalation is stopped & next lower dose is expanded to 12 patients to confirm the MTD.

SECONDARY OUTCOMES:
Pharmacokinetic parameters of C max , T max , AUC (tau), and t ½. | C 1 D 1 hrs 0, 1, 2, D 8 hrs 0, :15, :30, 1, 2, 4, 6, D 9 hrs 24, D 15 at hrs 0
  The secondary outcome measures of PKs, PDs, MMP7, hair follicle sampling, and Response Criteria by RECIST comprise the correlative studies of this trial and are designed to evaluate PK profiles, assess and evaluate the utility of potential biomarkers, and evaluate antineoplastic activity of PRI-724 + Gemcitabine.
Pharmacodynamic mRNA expression of survivin | C 1 D 1, D 8, D 15, D 22, All Cycles D 22, end of treatment
  The secondary outcome measures of PKs, PDs, MMP7, hair follicle sampling, and Response Criteria by RECIST comprise the correlative studies of this trial and are designed to evaluate PK profiles, assess and evaluate the utility of potential biomarkers, and evaluate antineoplastic activity of PRI-724 + Gemcitabine
Evaluation of antineoplastic activity of PRI-724 + gemcitabine per RECIST 1.1 criteria | Screening, end of C 2, every 2 cycles, end of treatment
  The secondary outcome measures of PKs, PDs, MMP7, hair follicle sampling, and Response Criteria by RECIST comprise the correlative studies of this trial and are designed to evaluate PK profiles, assess and evaluate the utility of potential biomarkers, and evaluate antineoplastic activity of PRI-724 + Gemcitabine
MMP7 levels in blood as ng/ml | C 1 Wk 1, Wk 4, Wk 4 all cycles, end of treatment
  The secondary outcome measures of PKs, PDs, MMP7, hair follicle sampling, and Response Criteria by RECIST comprise the correlative studies of this trial and are designed to evaluate PK profiles, assess and evaluate the utility of potential biomarkers, and evaluate antineoplastic activity of PRI-724 + Gemcitabine.
Gene expressions in hair follicle epithelial cells | Screening, C 1 D 14, C 2 Wk 4, end of treatment
  The secondary outcome measures of PKs, PDs, MMP7, hair follicle sampling, and Response Criteria by RECIST comprise the correlative studies of this trial and are designed to evaluate PK profiles, assess and evaluate the utility of potential biomarkers, and evaluate antineoplastic activity of PRI-724 + Gemcitabine

CONTACTS AND LOCATIONS:
Overall Officials: Robert R. McWilliams, M.D., Principal Investigator — Mayo Clinic
Locations (5):
- United States (5):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University of Washington Seattle Cancer Care Alliance, Seattle, Washington